CLINICAL TRIAL: NCT00664638
Title: Renal Denervation in Patients With Refractory Hypertension
Acronym: HTN-1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Vascular (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-037
Record Dates: First submitted 2008-04-21; First posted 2008-04-23 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Symplicty(TM) Catheter System — Renal denervation using the Symplicity Catheter System

SUMMARY:
To investigate the clinical utility of renal denervation in the treatment of refractory hypertension.

ELIGIBILITY:
Inclusion Criteria:

* >= 18 years of age
* a systolic blood pressure of 160mmHg or more
* receiving and adhering to full doses of at least three antihypertensive drugs
* estimated glomerular filtration rate (eGFR) of ≥45mL/min
* agrees to have the study procedure(s) performed and additional procedures and evaluations
* is competent and willing to provide written, informed consent to participate in this clinical study

Exclusion Criteria:

* hemodynamically or anatomically significant renal artery stenosis
* has a history or prior renal artery angioplasty
* has experienced MI, unstable angina pectoris, or CVA within 6 months
* has hemodynamically significant valvular heart disease
* has Type 1 diabetes
* has an implantable cardioverter defibrillator (ICD) or pacemaker, or any other metallic implant which is not compatible with magnetic resonance imaging (MRI)
* requires respiratory support
* is pregnant, nursing, or planning to be pregnant
* has known, unresolved history of drug use or alcohol dependency.
* is currently enrolled in another investigational drug or device trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2008-04; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
To document that renal denervation achieved via the delivery of RF energy is safe, and not associated with clinically significant adverse events, in patients with refractory hypertension. | 3 years

SECONDARY OUTCOMES:
To document the physiologic effects of renal denervation in patients with refractory hypertension. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Henry Krum, PhD, Principal Investigator — Monash University and The Alfred Hospital
Locations (9):
- Germany (9):
  - Herzzentrum Bad Krozingen, Bad Krozingen
  - St. Elisabeth Hospital, Bochum
  - Klinikum Coburg, Coburg
  - Universitaetsklinikum Duesseldorf, Düsseldorf
  - University of Erlangen at Nuremburg, Erlangen
  - CardioVascular Center Frankfurt, Sankt Katharinen, Frankfurt
  - Clinical Trial Center North, Hamburg
  - Universitatskliniken des Saarlandes, Homburg
  - University of Leipzig - Herzzentrum, Leipzig

REFERENCES:
- [Derived] Krum H, Schlaich MP, Sobotka PA, Bohm M, Mahfoud F, Rocha-Singh K, Katholi R, Esler MD. Percutaneous renal denervation in patients with treatment-resistant hypertension: final 3-year report of the Symplicity HTN-1 study. Lancet. 2014 Feb 15;383(9917):622-9. doi: 10.1016/S0140-6736(13)62192-3. Epub 2013 Nov 7. PMID 24210779
- [Derived] Mahfoud F, Ukena C, Schmieder RE, Cremers B, Rump LC, Vonend O, Weil J, Schmidt M, Hoppe UC, Zeller T, Bauer A, Ott C, Blessing E, Sobotka PA, Krum H, Schlaich M, Esler M, Bohm M. Ambulatory blood pressure changes after renal sympathetic denervation in patients with resistant hypertension. Circulation. 2013 Jul 9;128(2):132-40. doi: 10.1161/CIRCULATIONAHA.112.000949. Epub 2013 Jun 18. PMID 23780578
- [Derived] Mahfoud F, Schlaich M, Kindermann I, Ukena C, Cremers B, Brandt MC, Hoppe UC, Vonend O, Rump LC, Sobotka PA, Krum H, Esler M, Bohm M. Effect of renal sympathetic denervation on glucose metabolism in patients with resistant hypertension: a pilot study. Circulation. 2011 May 10;123(18):1940-6. doi: 10.1161/CIRCULATIONAHA.110.991869. Epub 2011 Apr 25. PMID 21518978
- [Derived] Krum H, Schlaich M, Whitbourn R, Sobotka PA, Sadowski J, Bartus K, Kapelak B, Walton A, Sievert H, Thambar S, Abraham WT, Esler M. Catheter-based renal sympathetic denervation for resistant hypertension: a multicentre safety and proof-of-principle cohort study. Lancet. 2009 Apr 11;373(9671):1275-81. doi: 10.1016/S0140-6736(09)60566-3. Epub 2009 Mar 28. PMID 19332353